CLINICAL TRIAL: NCT00095641
Title: S0225: Phase II Study of Adjuvant Low-Dose Capecitabine After Salvage Surgery in Patients With Locally Recurrent or Persistent Squamous Cell Carcinoma of the Head and Neck
Brief Title: S0225 Capecitabine in Treating Patients Who Have Undergone Surgery for Locally Recurrent or Persistent Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no longer studying this disease site
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000394169; S0225 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Capecitabine; Chemotherapy, Adjuvant; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Procedure: adjuvant therapy
Procedure: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving capecitabine after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well capecitabine works in treating patients who have undergone surgery for locally recurrent or persistenthead and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine 2-year disease-free survival of patients treated with surgical salvage followed by adjuvant low-dose capecitabine for locally recurrent or persistent squamous cell carcinoma of the head and neck .
* Determine the toxic effects of this drug in these patients.
* Determine 2-year overall survival of patients treated with this drug.
* Determine patterns of disease relapse in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine once daily for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck
* Locoregionally recurrent or persistent disease
* No thyroid gland, salivary gland, or nasopharynx disease sites
* Must have undergone definitive or post-operative radiotherapy at the time of initial curative treatment
* Must have undergone salvage surgical resection within the past 56 days
* All current disease must be completely resected, including resection of recurrent primary disease and/or neck dissection, if regional nodal disease is present
* Surgical margins must be free of disease on final pathological evaluation of specimens
* No definitive or adjuvant radiotherapy or reirradiation for recurrent or persistent disease allowed at the time of salvage treatment
* No evidence of distant disease by clinical examination and CT scan of the chest and upper abdomen (including the liver) within the past 90 days

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine clearance ≥ 30 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to take oral tablets OR able to take crushed tablets through a gastrostomy tube
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy
* No concurrent filgrastim (G-CSF)

Chemotherapy

* Prior systemic chemotherapy as definitive therapy for head and neck cancer allowed (prior treatment with fluorouracil allowed, but must be catalogued)
* More than 5 years since prior systemic chemotherapy for any other cancer diagnosis
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy
* Concurrent hormonal therapy for non-cancer diagnosis allowed

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schwartz, MD, Study Chair — M.D. Anderson Cancer Center